CLINICAL TRIAL: NCT02248519
Title: Laparoscopic Versus Open Gastrectomy for Gastric Cancer, a Multicenter Prospectively Randomized Controlled Trial (LOGICA-trial)
Brief Title: Laparoscopic Versus Open Gastrectomy for Gastric Cancer
Acronym: LOGICA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Richard van Hillegersberg, MD PhD, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL47444.041.14
Record Dates: First submitted 2014-09-17; First posted 2014-09-25 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Gastrectomy; Laparoscopy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open Gastrectomy (Active Comparator): Patients allocated to the 'Open Gastrectomy' group will receive distal or total gastrectomy via laparotomy. This group is considered the control group
  Interventions: Procedure: Open Gastrectomy
- Laparoscopic Gastrectomy (Experimental): Patients allocated to the 'Laparoscopic Gastrectomy' group will undergo distal or total gastrectomy via laparoscopy.
  Interventions: Procedure: Laparoscopic Gastrectomy

INTERVENTIONS:
Procedure: Open Gastrectomy — Patients allocated to the 'Open Gastrectomy' group will receive distal or total gastrectomy via laparotomy. This group is considered the control group
  Arms: Open Gastrectomy
Procedure: Laparoscopic Gastrectomy — Patients allocated to the 'Laparoscopic Gastrectomy' group will undergo distal or total gastrectomy via laparoscopy. If laparoscopic resection does not seem feasible during surgery, the procedure may be converted to an open gastrectomy.
  Arms: Laparoscopic Gastrectomy

SUMMARY:
This is the first randomized controlled trial comparing laparoscopic and open gastrectomy for resectable gastric cancer in a Western population. The hypothesis is that laparoscopic gastrectomy will result in a lower post-operative burden by means of shorter post-operative hospital stay. Secondarily that laparoscopic gastrectomy is hypothesized to be associated with lower post-operative morbidity and readmissions, higher cost-effectiveness, and better post-operative quality of life, with similar mortality and oncologic outcomes, compared to open gastrectomy. The study starts on 1 December 2014. Inclusion and follow-up will take three and five years respectively. Short-term results will be analyzed and published after discharge of the last randomized patient.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the stomach
* Surgically resectable (cT1-4a, N0-3b, M0) tumor
* Age ≥ 18 years
* European Clinical Oncology Group (ECOG) performance status 0, 1 or 2.
* Written informed consent

Exclusion Criteria:

* Siewert type I esophagogastric junction tumor
* Non-elective surgery
* Previous gastric resection or recurrent gastric cancer
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative hospital stay | During admission, an expected average of 2 weeks
  The primary outcome of this study is the post-operative hospital stay (days), since this is considered a strong end point as it reflects the impact of the different surgical procedures.

SECONDARY OUTCOMES:
Mortality | 30 days post-operative
  Measured as 30-day mortality rate
Post-operative morbidity | Up to 5 years post-operative
  Complications will be classified according to the Clavien-Dindo system and include anastomotic leakage, anastomotic stricture, respiratory complications, cardiac complications, intra-abdominal bleeding , intra-abdominal abscess, sepsis, ileus, wound infection, fistula, urinary tract infection and dumping syndrome
Cost-effectiveness | Up to 5 years post-operative
  Cost-effectiveness will be calculated by comparing the direct medical cost related to both strategies up until five years after the operation
Quality of Life | Up to 5 years post-operative
  The validated quality of life questionnaires EORTC QLQ-30, EORTC QLQ-STO22 and EQ-5D-5L, will be filled in pre-operative <5 days and post-operative at 6 weeks, 12, 24, 36, 48 and 60 months after surgery.
Readmissions | Up to 5 years post-operative
  The number of post-operative readmissions
Oncologic outcomes (R0-resection rate and lymph node yield) | Pathology report 1-2 weeks after surgery
  R0-resection rate of the distal and proximal margin, defined according to the College of American Pathologists. Lymph node yield: the amount of harvested lymph nodes per patient.

OTHER OUTCOMES:
Perioperative blood loss | Post-operative day 1
  Measured in milliliters (ml)
Operative time | Post-operative day 1
  The time from incision to closure of all wounds in minutes (min)
Conversion rate | Post-operative day 1
  The percentage (%) of laparoscopic gastrectomies that had to be converted intra-operatively to an open procedure due to any reason.
Survival | Up to 5 years post-operative
  Measured as 5-year disease free survival and 5-year overall survival
VAS-score | Post-operative day 1 and 2
Surgeons ergonomics | Post-operative day 1
  Measured with the Subjective Mental Effort Questionnaire (SMEQ)
Time to return to normal nutritional regime | Up to 5 years post-operative
Time to return to daily activity | Up to 5 years post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Richard van Hillegersberg, MD PhD, Principal Investigator — Dept. of Surgery, University Medical Center Utrecht
Locations (10):
- Netherlands (10):
  - Zorggroep Twente Almelo, Almelo
  - Meander Medical Center, Amersfoort
  - VU University Medical Center, Amsterdam
  - Academic Medical Center, Amsterdam
  - Gelre Hospital, Apeldoorn
  - Catharina Hospital, Eindhoven
  - Leiden University Medical Center, Leiden
  - Erasmus Medical Center, Rotterdam
  - Zuyderland Medical Center, Sittard-Geleen
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary manuscript will be shared after de-identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Immediately following publication; no end date.
Access Criteria: Anyone who wishes to access the data for any purpose.

REFERENCES:
- [Background] Haverkamp L, Brenkman HJ, Seesing MF, Gisbertz SS, van Berge Henegouwen MI, Luyer MD, Nieuwenhuijzen GA, Wijnhoven BP, van Lanschot JJ, de Steur WO, Hartgrink HH, Stoot JH, Hulsewe KW, Spillenaar Bilgen EJ, Rutter JE, Kouwenhoven EA, van Det MJ, van der Peet DL, Daams F, Draaisma WA, Broeders IA, van Stel HF, Lacle MM, Ruurda JP, van Hillegersberg R; LOGICA study group. Laparoscopic versus open gastrectomy for gastric cancer, a multicenter prospectively randomized controlled trial (LOGICA-trial). BMC Cancer. 2015 Jul 29;15:556. doi: 10.1186/s12885-015-1551-z. PMID 26219670
- [Derived] van der Veen A, Ramaekers M, Marsman M, Brenkman HJF, Seesing MFJ, Luyer MDP, Nieuwenhuijzen GAP, Stoot JHMB, Tegels JJW, Wijnhoven BPL, de Steur WO, Kouwenhoven EA, Wassenaar EB, Draaisma WA, Gisbertz SS, van der Peet DL, May AM, Ruurda JP, van Hillegersberg R; LOGICA study group. Pain and Opioid Consumption After Laparoscopic Versus Open Gastrectomy for Gastric Cancer: A Secondary Analysis of a Multicenter Randomized Clinical Trial (LOGICA-Trial). J Gastrointest Surg. 2023 Oct;27(10):2057-2067. doi: 10.1007/s11605-023-05728-3. Epub 2023 Jul 18. PMID 37464143
- [Derived] de Jongh C, van der Veen A, Brosens LAA, Nieuwenhuijzen GAP, Stoot JHMB, Ruurda JP, van Hillegersberg R; LOGICA Study Group. Distal Versus Total D2-Gastrectomy for Gastric Cancer: a Secondary Analysis of Surgical and Oncological Outcomes Including Quality of Life in the Multicenter Randomized LOGICA-Trial. J Gastrointest Surg. 2023 Sep;27(9):1812-1824. doi: 10.1007/s11605-023-05683-z. Epub 2023 Jun 20. PMID 37340107
- [Derived] van der Veen A, Brenkman HJF, Seesing MFJ, Haverkamp L, Luyer MDP, Nieuwenhuijzen GAP, Stoot JHMB, Tegels JJW, Wijnhoven BPL, Lagarde SM, de Steur WO, Hartgrink HH, Kouwenhoven EA, Wassenaar EB, Draaisma WA, Gisbertz SS, van der Peet DL, May AM, Ruurda JP, van Hillegersberg R; LOGICA Study Group. Laparoscopic Versus Open Gastrectomy for Gastric Cancer (LOGICA): A Multicenter Randomized Clinical Trial. J Clin Oncol. 2021 Mar 20;39(9):978-989. doi: 10.1200/JCO.20.01540. Epub 2021 Jan 6. PMID 34581617